CLINICAL TRIAL: NCT00498459
Title: Intervention Centered on Adolescents' Physical Activity and Sedentary Behavior (ICAPS)
Acronym: ICAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louis Pasteur University, Strasbourg (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other); National Nutritional Health Program, France (Other); Minister of Youth Affairs and Sports, France (Other Government)
Responsible Party: Principal Investigator, Chantal Simon, Professor, Louis Pasteur University, Strasbourg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2007_01
Record Dates: First submitted 2007-07-09; First posted 2007-07-10 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Physical Activity; Overweight; Cardiovascular Disease
Keywords: Physical activity; Randomised trial; Prevention; Adolescents; Obesity; Cardiovascular risk factors
MeSH Terms: conditions — Motor Activity; Overweight; Cardiovascular Diseases; Obesity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ICAPS (Experimental): Promotion Physical Activity
  Interventions: Behavioral: Physical activity
- Control (No Intervention): No specific physical activity promotion Ususal school program

INTERVENTIONS:
Behavioral: Physical activity — Physical promotion according to socio-ecological model Limitation of sedentary behaviour
  Arms: ICAPS

SUMMARY:
Physical activity is thought to be a key element in preventing the obesity epidemic and the associated cardiovascular and metabolic diseases. However population-based studies directed at promoting physical activity in youth have shown limited success in obesity prevention. The aim of this study is to assess whether an intervention integrating socioecological changes, which has the potential to induce sustained changes in physical activity, prevents overweight and cardiovascular risk in adolescents.

DETAILED DESCRIPTION:
Background

Physical activity is thought to be a key element in preventing the obesity epidemic and the associated cardiovascular and metabolic diseases. However population-based studies directed at promoting physical activity in youth have shown limited success in obesity prevention. The aim of this study is to assess whether an intervention integrating socioecological changes, which has the potential to induce sustained changes in physical activity, prevents overweight and cardiovascular risk in adolescents.

Methods

Population and design: The Intervention Centered on Adolescents' Physical activity and Sedentary behavior (ICAPS) is a 4-year randomized prevention study targeting 6th graders (e.g. 12 year old adolescents). The study design is based on a randomization at school level and follows the intention-to-treat principle. Eight schools (four intervention schools and four controls) are randomly selected out of the 77 public middle schools of the Department of Bas-Rhin (Eastern France). To balance potential confounding factors and to ensure a broad socioeconomic context, randomization is done after stratification on sociogeographical criteria. Intervention status of the schools is randomized in each pair of matched schools. All initially first-level students of the randomized schools are eligible to participate.

Intervention: The 4-year intervention program is designed to promote physical activity by changing attitudes through debates and access to attractive activities, and by providing social support and environmental changes encouraging physical activity. The students of the control schools follow their usual school curriculum and physical education classes and are not be submitted to any intervention.

Outcomes and follow-up: The primary outcome is the subjects' body mass index (BMI). Prespecified secondary end points include body composition, physical activity and sedentary behaviors, attitudes towards physical activity, and various cardiovascular risk factors. Surveys take place at baseline and annually at the end of each school year. Fasting blood is sampled at baseline and every two years. Physical examinations are performed by qualified professionals and questionnaires are administered to small groups of 3 to 6 students. All the procedures are standardized among schools and the interviewers are be regularly trained to assure the reliability of the measurements.

Statistical analysis: Outcome data are analyzed using mixed linear models taking into account the cluster randomization design and the repeated individual data. Random effects are schools within intervention group and individuals within schools. Possible heterogeneity of the intervention's effect according to gender and initial weight status will be tested.

Perspectives This study will assess the feasibility and the efficacy of a multilevel multipartnership prevention program targeting adolescents' physical activity.

ELIGIBILITY:
Inclusion Criteria:

* 6th graders (in 2002)
* student in one of the eight randomised middle school (four pairs of middle-school located in Bas-Rhin, France)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 954 (Actual)
Dates: Start 2002-09; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
body-mass index | at the end of the second, third and fourth school years of intervention

SECONDARY OUTCOMES:
fat mass (impedancemetry) | at the end of the second, third and fourth school years of intervention
physical activity (MOSPA) | at the end of the second, third and fourth school years of intervention
Attitudes and motivation toward physical activity | at the end of the second, third and fourth school years of intervention
clinical and biological cardiovascular risk factors | at the end of the second, and fourth school years of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Chantal Simon, PhD, MD, Study Chair — Louis Pasteur University of Strasbourg
Locations (1):
- Louis Pasteur University of Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No